CLINICAL TRIAL: NCT04767685
Title: The Bern Perioperative Biobank to Define Perioperative Changes of Molecular Markers of Perioperative Organo-dysfunctions, Inflammation, Adverse Events and Disease Progression
Brief Title: The Bern Perioperative Biobank
Acronym: BPBB
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09f
Record Dates: First submitted 2020-12-16; First posted 2021-02-23 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Surgical Procedure, Operative
Keywords: Genetic association study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood (plasma and cells)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Consenting patients undergoing non-emergency surgery with anesthesia

SUMMARY:
The goal of the research is to define clinically relevant molecular markers for increased risk of peri-/ postoperative organo-dysfunctions, inflammation, adverse events and disease progression. To better understand the perioperative impact the investigators aim to determine perioperative levels of molecular markers over time in the available samples and clinical data of the Bern perioperative Biobank (BPBB) cohort to finally increase quality of perioperative care of patients by permitting preventive measures to be taken early in patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Non-emergency surgery

Exclusion Criteria

* Transient incapacity to consent or insufficient time (< 6h) to consider study participation
* No informed consent
* Cognitive impairment/Patients unable to consent
* Patients who retrospectively expressed their wish to be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Assessing the change of the metabolic profile in the perioperative setting | Before induction of anesthesia as baseline
  Surgery causes significant disruption of physiologic metabolism. The investigators currently lack specific markers to assess change of the metabolic profile in the perioperative setting. The investigators aim to identify metabolic markers and their change in the perioperative period in association with patients' clinical outcome.
Assessing the change of the metabolic profile in the perioperative setting | Ca. 2-5hours later upon finishing the surgery
  Surgery causes significant disruption of physiologic metabolism. The investigators currently lack specific markers to assess change of the metabolic profile in the perioperative setting. The investigators aim to identify metabolic markers and their change in the perioperative period in association with patients' clinical outcome.
Assessing the change of the metabolic profile in the perioperative setting | On postoperative day 1 during the morning round between 07:30-9:00am
  Surgery causes significant disruption of physiologic metabolism. The investigators currently lack specific markers to assess change of the metabolic profile in the perioperative setting. The investigators aim to identify metabolic markers and their change in the perioperative period in association with patients' clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stüber, Prof. MD, Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern; Markus M Lüdi, MD, Study Director — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Bello C, Filipovic MG, Huber M, Flannery S, Kobel B, Fischer R, Kessler BM, Raber L, Stueber F, Luedi MM. Discovery of plasma proteome markers associated with clinical outcome and immunological stress after cardiac surgery. Front Cardiovasc Med. 2023 Dec 22;10:1287724. doi: 10.3389/fcvm.2023.1287724. eCollection 2023. PMID 38379859
- [Derived] Heinisch PP, Mihalj M, Huber M, Schefold JC, Hartmann A, Walter M, Steinhagen-Thiessen E, Schmidli J, Stuber F, Raber L, Luedi MM. Impact of Lipoprotein(a) Levels on Perioperative Outcomes in Cardiac Surgery. Cells. 2021 Oct 21;10(11):2829. doi: 10.3390/cells10112829. PMID 34831051